CLINICAL TRIAL: NCT03602352
Title: A Cohort Study of the Cost for Patients Operated for Adhesive Obstruction (SBO) During a Five-year Period
Brief Title: A Study of the Cost for Patients Operated for Adhesive Obstruction (SBO) During a Five-year Period
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: ASBO-02
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Adhesive Small Bowel Obstruction
Keywords: Cohort; Surgery; Adhesive Small Bowel Obstruction; Cost

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cohort study of the cost for patients operated for adhesive small bowel obstruction (SBO) during a five-year period

DETAILED DESCRIPTION:
It is a population-based cohort study of the costs for patients operated for adhesive small bowel obstruction during a five-year period (2007-2012) in two Swedish neighboring regions. Patients were identified by a broad search of operation and International Classification of Diseases (ICD) codes. Data regarding surgery and complications has been analyzed in a previous study (Clinical trials no NCT0353459)

The costs for hospital stay, radiology, Intensive Care Unit (ICU)-care, operation for the index SBO care event were calculated. The cost for revisit, sick leave and recurrent SBO during follow-up were calculated. Patients were followed to 31st January 2017, last medical note or death.

ELIGIBILITY:
Inclusion Criteria:

* Above18 years of age
* Surgery for adhesive surgical bowel obstruction (SBO)

Exclusion Criteria:

• Surgery for SBO of other etiology than adhesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery due to adhesive small bowel obstructions during the time period 2007-2012.
Sampling Method: Non-Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Cost for primary hospital admission in patients who underwent SBO surgery during 2007-2012 | 2007-2012
  Per 100 000 inhabitants and year

SECONDARY OUTCOMES:
Cost for further hospital admissions, surgery and outpatient visits during follow-up | 2007-2012
Potential cost-reduction with prophylactic treatment calculating with different prophylactic efficacy levels | 2007-2012

CONTACTS AND LOCATIONS:
Overall Officials: Urban Karlbom, MD PhD, Study Chair — Region Uppsala